CLINICAL TRIAL: NCT02063295
Title: Randomized, Double-Blind, Placebo Controlled, Phase 2a Trial of ZGN-440 (Subcutaneous Beloranib in Suspension), A Novel Methionine Aminopeptidase 2 Inhibitor, in Obese Subjects With Hypothalamic Injury to Evaluate Weight Reduction and Safety Over 4 Weeks Followed by an Optional 4-Week Open-Label Extension
Brief Title: An Efficacy, Safety, and Pharmacokinetics Study of Beloranib in Obese Subjects With Hypothalamic Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZAF-221
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Over-weight; Hypothalamic Injury; Craniopharyngioma
Keywords: Beloranib; ZGN-440; ZGN-440 for injectable suspension; ZGN-433
MeSH Terms: conditions — Obesity; Craniopharyngioma | interventions — CKD732

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZGN-440 sterile diluent (Placebo Comparator): Subjects will receive placebo twice weekly subcutaneous injections for 4 weeks.
  Interventions: Drug: ZGN-440 sterile diluent
- ZGN-440 for injectable suspension (Experimental): Subjects will receive ZGN-440 for injectable suspension (beloranib) twice weekly subcutaneous injections for up to 8 weeks.
  Interventions: Drug: ZGN-440 for injectable suspension

INTERVENTIONS:
Drug: ZGN-440 sterile diluent — ZGN-440 sterile diluent/placebo
  Other Names: Placebo
  Arms: ZGN-440 sterile diluent
Drug: ZGN-440 for injectable suspension
  Other Names: ZGN-440; Beloranib
  Arms: ZGN-440 for injectable suspension

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of beloranib in obese subjects with hypothalamic injury.

ELIGIBILITY:
Inclusion Criteria:

* Obesity as a consequence of acquired anatomical hypothalamic damage as evidenced by BMI ≥30 and ≤60 kg/m2
* Greater than 6 months post-treatment, including chemotherapy, surgery or radiation with resulting injury to the hypothalamus and/or the pituitary
* Stable body weight for at least 3 months
* Type 2 diabetes mellitus is allowed

Exclusion Criteria:

* Males taking gonadotropin replacement therapy (LH/FSH)
* Subjects who are planning any fertility treatment within 6 months of study participation
* Use of weight loss agents, including herbal medications, in the past 3 months
* Current or anticipated chronic use of narcotics or opiates
* History of severe psychiatric disorders
* Type 1 diabetes mellitus
* Metabolic disorders or genetic disorders linked to obesity
* History of any bariatric surgery
* Participation in any clinical study with an investigational drug or device within the 3 months prior to enrollment in this study
* Blood loss or donation >500 mL within the past 3 months
* Females who are pregnant, nursing, intend to become pregnant during the study or any males who plan to father/conceive a child within 6 months after completion of study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline to the end of the randomized dosing period. | 4 weeks

SECONDARY OUTCOMES:
Change in lipid profile (cholesterol, LDL, HDL, triglycerides) from baseline to the end of the randomized dosing period | 4 weeks
Change in hs-CRP from baseline to the end of the randomized dosing period. | 4 weeks
Change in hunger from baseline to the end of the randomized dosing period. | 4 weeks
Change in quality of life from baseline to the end of the randomized dosing period. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (2):
  - The Boden Institute, Sydney, New South Wales
  - Austin Health, Metabolic Disorders Centre, Heidelberg Heights, Victoria

REFERENCES:
- [Derived] Shoemaker A, Proietto J, Abuzzahab MJ, Markovic T, Malloy J, Kim DD. A randomized, placebo-controlled trial of beloranib for the treatment of hypothalamic injury-associated obesity. Diabetes Obes Metab. 2017 Aug;19(8):1165-1170. doi: 10.1111/dom.12928. Epub 2017 Apr 18. PMID 28261955